CLINICAL TRIAL: NCT04415775
Title: Changes in Metabolic Activity, and Gait Function by Dual-task Cognitive Game-based Treadmill Intervention in Parkinson's Disease
Acronym: CMAGDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Weston Brain Institute (Other)
Responsible Party: Principal Investigator, Dr. Tony Szturm, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B2020:043
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
Keywords: Dual task walking; Treadmill walking; PET scans; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: One experimental group and other control group receiving control intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual-task walking Intervention (Experimental)
  Interventions: Other: Game based treadmill Program
- Conventional Gait Rehabilitation (Active Comparator)
  Interventions: Other: Conventional Gait Rehabilitation
- Healthy Controls (No Intervention)

INTERVENTIONS:
Other: Game based treadmill Program — Participants will be expected to play several cognitive computer games while standing on a sponge pad (10-min warm-up and while walking on the treadmill at your self-selected comfortable speed. (Dual-task treadmill training). This would be done in intervals of 2-4 min with rest periods for a total time of 35 minutes Treadmill speed and the difficulty level of the cognitive games will progress depending on participant performance and comfort level.
  Arms: Dual-task walking Intervention
Other: Conventional Gait Rehabilitation — Participants will undergo a mixture of current gait training programs available for people with Parkinson's Disease. The protocol will be a Warm-up exercise consisting of rhythmical large movements (10 minutes), as well as video game practice while standing (i.e., single-task; 10 minutes). Treadmill walking in intervals of 2-4 minutes with rest periods. Walking over the ground while negotiating through obstacles. (10 minutes) The speed of the treadmill will be progressed gradually and as tolerated.
  Arms: Conventional Gait Rehabilitation

SUMMARY:
The present proposal will evaluate the neural underpinnings of (a) the decline of mobility function in Parkinson's disease (PD), and (b) the effects of an innovative computer-guided dual-task (DT) mobility training platform (complementary approach: exercise intervention). Improved mobility functioning in PD, specifically balance, gait and cognition, directly translates to improved community ambulation as well as increased physical activity and social participation. These benefits are known to have a significant preventive and disease-modifying impact that surpasses any currently available pharmacological interventions. Outcomes of this research will provide new insights into brain plasticity mechanisms and will accelerate further optimization and commercialization of multi-modal mobility-cognitive training applications along with accompanying smart electronic monitoring tools. With wider usage of this training platform, rehabilitation specialists will be able to effectively scale services, while still monitoring quality and ensuring accountability. Thus, the study is highly transformative.

DETAILED DESCRIPTION:
The present proposal will evaluate the neural underpinnings of (a) the decline of mobility function in Parkinson's disease (PD), and (b) the effects of an innovative computer-guided dual-task (DT) mobility training platform (complementary approach: exercise intervention). Improved mobility functioning in PD, specifically balance, gait and cognition, directly translates to improved community ambulation as well as increased physical activity and social participation. These benefits are known to have a significant preventive and disease-modifying impact that surpasses any currently available pharmacological interventions. Outcomes of this research will provide new insights into brain plasticity mechanisms and will accelerate further optimization and commercialization of multi-modal mobility-cognitive training applications along with accompanying smart electronic monitoring tools. With wider usage of this training platform, rehabilitation specialists will be able to effectively scale services, while still monitoring quality and ensuring accountability. Thus, the study is highly transformative.

The investigators propose a collaborative project between our research centers at the University of Manitoba and the University of Toronto, to further understand the neural underpinnings of cognition/gait impairment and the effects of DT training in PD.

Cutting-edge behavioural brain imaging methods will be used to identify functional brain metabolic network re-organization and the molecular basis of gait/cognitive impairment. This will be used to evaluate the neurophysiological underpinnings of the DT treadmill training effect, which has repeatedly demonstrated to be clinically effective. The possibility of detecting these changes and localizing the site(s) of brain plasticity will have important implications at several levels. These biomarkers could be used as an indicator of disease severity, outcome measures for neuroprotection studies and other treatment and lifestyle strategies.

Objective 1: To characterize the abnormal brain metabolic pattern in PD patients during DT-walking as compared to healthy age-matched controls.

Objective 2: The investigators will examine whether a 10-week treadmill walking program combined with specific cognitive activities (i.e. true DT walking training known to improve gait function and reduce falls) will "normalize" the brain abnormality (that is identified in Aim 1), or whether it will activate a novel compensatory mechanism and therefore evidence to isolate the region(s) of brain plasticity.

The hypothesis is that the DT gait-related abnormal brain metabolic pattern and abnormally elevated amyloid deposition are inter-related and that these abnormal functional connectivity patterns and structural changes are highly associated with gait, cognitive and DT walking deficits in PD. It is also hypothesized that the DT treadmill-training program will result in specific and significant changes in the DT gait-related abnormal brain metabolic pattern, in the PD participants.

ELIGIBILITY:
Inclusion Criteria: (PD Participants)

* Diagnosed with idiopathic PD, defined by the UK Brain Bank criterion in disease stage 2 - 3 (classified by Hoehn and Yahr scale),
* Montreal cognitive assessment (MoCA) scores to be 25 or higher
* Age 55-70 years
* Stable medications for Parkinson over the past 3 months
* Able to walk at least 50m without any assistive device
* Episode of FOG in the past 6 months

Exclusion Criteria: (PD Participants)

* The presence of neurological conditions other than PD affecting cognitive abilities.
* Any orthopedic impairment affecting gait and balance.
* Any cardiovascular impairment limiting the ability to walk for 10-15 minutes on a treadmill;
* Abnormal MRI
* General contraindications.

Inclusion Criteria: (Healthy Controls)

* Age 55-70 years,
* Independent community living,
* Not receiving any home care or Physiotherapy,
* Walking outdoors for exercise for at least 3 times per week,
* No neurological conditions affecting mobility or affecting cognitive abilities,
* Any orthopedic impairment affecting gait and balance.
* Any cardiovascular impairment limiting the ability to walk for 10-15 minutes on a treadmill.
* Abnormal MRI and
* General contraindications for PET and MRI including severe dyskinesia, diabetes, cardiac pacemakers.

Exclusion Criteria (Healthy Controls):

* Any orthopedic impairment affecting gait and balance.
* Any cardiovascular impairment limiting the ability to walk for 10-15 minutes on a treadmill.
* Abnormal MRI
* General contraindications.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
NDWP scores | 10 weeks
  NDWP scores on PET scans of participants will be analysed to identify gait impairment related imagining signatures during single and dual-task walking, and after intervention. They will also be compared to age-matched healthy controls using student t-test.
Step Length Coefficient of Variability | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- College of Rehabilitation Sciences, University of Manitoba, Winnipeg, Manitoba, Canada